CLINICAL TRIAL: NCT02857452
Title: Transcultural Validation in French of the Systemic Lupus Activity Questionnaire (SLAQ) and the Lupus Quality Of Life (LupusQoL) Questionnaire
Acronym: FRESH COLA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: DEVILLIERS 189 HORS AOI 2008
Record Dates: First submitted 2016-08-02; First posted 2016-08-05 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-07

CONDITIONS: Lupus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Lupus
  Interventions: Other: SLA Questionnaire; Other: Lupus Qol Questionnaire

INTERVENTIONS:
Other: SLA Questionnaire
Other: Lupus Qol Questionnaire

SUMMARY:
The evaluation of lupus patients must include several approaches, in particular disease activity and quality of life.

The Systemic Lupus Activity Questionnaire (SLAQ) is a validated self-questionnaire to evaluate disease activity. It has the advantage of being inexpensive, easy to use in large cohorts and has been used in several studies. It has never been validated in French. The Lupus Quality Of Life (LupusQoL) is a self-questionnaire to evaluate quality of life and is specific to systemic lupus erythematous; it was developed from interviews with patients.

This tool, validated in a British population, has never been validated in French.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lupus meeting the 1997 classification criteria of the American College of Rheumatology for systemic lupus erythematous.
* Patients able to understand written and spoken French.
* Patients who have been informed about the research

Exclusion Criteria:

* Severe mental retardation.
* Any impairment of ability to understand making self-evaluation impossible.
* Age < 18 years.
* Age > 75 years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lupus meeting the 1997 classification criteria of the American College of Rheumatology for systemic lupus erythematous
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2009-01; Primary Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Answers in French to the au Systemic Lupus Activity Questionnaire (SLAQ) | Evolution of answers between D0, D15, M3 and M6

SECONDARY OUTCOMES:
Answers in French to the Lupus Quality of Life (Lupus QoL) questionnaire | Evolution of answers between D0, D15, M3 and M6

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France